CLINICAL TRIAL: NCT04768101
Title: Quantitative Imaging of Brain Glymphatic Function in Humans
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Manus Donahue, Professor of Neurology, Psychiatry and Behavioral Sciences, and Radiology and Radiological Sciences, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Imaging of Brain Glymphatics
Record Dates: First submitted 2021-02-16; First posted 2021-02-24 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Intervention Model Description: There is no masking in this protocol.
Masking Description: There is no masking in this protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson's Disease participants with MCI (Experimental): Patient volunteers will also undergo a C-11 PiB PET scan. This procedure utilizes a common radiotracer that is used routinely in clinical PET scans and will be purchased here from PETNET and certified for human use. All PET scans will be performed by a certified PET technologist at the Vanderbilt University Institute of Imaging Science.
  Interventions: Drug: [11C]-PIB

INTERVENTIONS:
Drug: [11C]-PIB — [11C]-PIB is a PET radiotracer used to evaluate levels of Αβ burden.
  Other Names: N-Methyl-[ 11C]-2-(4'-methylaminophenyl)-6-hydroxybenzothiasole; [11C]-Pittsburgh Compound B; [ 11C]6-OH-BTA-1

SUMMARY:
Recent immunological and physiological studies have provided evidence in support of a central nervous system (CNS) lymphatic drainage system in vertebrate animals, and preliminary evidence has suggested that a similar system exists in humans. If operative, this system may have central relevance to many vascular and fluid clearance disorders such as stroke, multiple sclerosis, Parkinson's disease, and Alzheimer's disease related dementia (ADRD): diseases which represent some of the most pressing healthcare challenges of the 21st century. Evaluating this possibility will require improved, robust imaging methods sensitive to lymphatic drainage dysfunction; as such, the goal of this work is to apply novel magnetic resonance imaging approaches, optimized already for evaluating lymphatic circulation in patients with peripheral lymphatic dysfunction, to quantify relationships between physiological hallmarks of ADRD and CNS lymphatic function in humans.

DETAILED DESCRIPTION:
The proposal involves magnetic resonance imaging (MRI) of healthy volunteers and patient volunteers suffering from Parkinson's disease. As part of the research study, volunteers will undergo 1-2 non-invasive MRI scans at a field strength of 3 Tesla. Each scan session will last 60-90 minutes, and will include the time when the volunteers will rehearse the experiment outside of the scanner, time for the volunteers and patients to be comfortably placed in the scanner, scanning, and finally time for the patients to slowly exit the scan room.

All MRI methods are non-invasive and no exogenous contrast agents will be required.

Patient volunteers will also undergo an C-11 PiB PET scan for Aim (2). This procedure utilizes a common radiotracer that is used routinely in clinical PET scans and will be purchased here from PETNET and certified for human use. All PET scans will be performed by a certified PET technologist at the Vanderbilt University Institute of Imaging Science.

Finally, in Aim (3) of this study, measurements of glymphatic function will be performed before and during general anesthesia. Importantly, the general anesthesia will be administered as part of standard-of-care for clinically-indicated MRIs required for deep brain stimulation planning and electrode placement. Therefore, the intervention itself is not a research procedure. Additionally, the scan that will be performed, which is a modified diffusion tensor imaging (DTI) MRI approach, is already performed as part of this clinical protocol. Therefore, it is anticipated that the participant will not be sedated any longer than what would be required for clinical indication for this procedure. As such, while this study qualifies as a clinical trial by NIH criteria, it is expected to pose no more risk than what the participant will receive from their clinical standard-of-care procedure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's Disease or controls
* willing to participate in PET and MRI imaging

Exclusion Criteria:

* recent stimulant use
* unstable diabetes
* prior stroke
* claustrophobia
* prior cancer treatment with chemotherapy
* history of traumatic brain injury
* any unstable medical condition

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diffusion Tensor Imaging Along Perivascular Spaces (DTI-ALPS) | baseline, under anesthesia
  Using a 3T MRI (body coil transmission and SENSE phased-array 32-channel reception), images will be taken. For analysis, a unitless ratio of diffusion along perivascular space relative to orthogonal to perivascular space at the level of the lateral brain ventricles will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Manus J Donahue, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data may be shared upon request by other researchers.
Supporting Information: SAP, CSR
Time Frame: upon request
Access Criteria: upon request